CLINICAL TRIAL: NCT03251001
Title: Acellular Dermal Matrix Allograft Versus Free Gingival Graft: a Histological Evaluation and Split-mouth Randomized Clinical Trial
Brief Title: Acellular Dermal Matrix Allograft Versus Free Gingival Graft
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Carla Andreotti Damante, Associate professor, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BauruSchoolDentistryADM
Record Dates: First submitted 2017-08-09; First posted 2017-08-16 (Actual); Last update posted 2018-03-09 (Actual); Status verified 2018-03

CONDITIONS: Gingiva Atrophy; Gingivitis
Keywords: gingiva; keratinized mucosa; gingival graft
MeSH Terms: conditions — Gingival Recession; Gingivitis | interventions — Transplantation, Homologous

STUDY DESIGN:
Intervention Model Description: Split-mouth design. One side of mouth was test group, other side was control group.
Who Masked: Outcomes Assessor
Masking Description: All clinical parameters were evaluated by a calibrated examiner (intraclass correlation coefficient = 0.98) blind to test and control groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Control (Active Comparator): Sites receiving a free gingival graft
  Interventions: Procedure: Control
- Device - Acellular dermal matrix (Experimental): Sites receiving acellular dermal matrix
  Interventions: Device: Acellular Dermal Matrix

INTERVENTIONS:
Procedure: Control — Free epithelized gingival graft, harvested from palate, was grafted in a site with lack of keratinized gingiva
  Arms: Control
Device: Acellular Dermal Matrix — Acellular Dermal Matrix was grafted in a site with lack of keratinized gingiva, in substitution of an autogenous graft from patient palate
  Other Names: allograft
  Arms: Device - Acellular dermal matrix

SUMMARY:
The present split-mouth controlled randomized clinical trial aimed to evaluate clinical and histological results of acellular dermal matrix allograft (ADM) compared to autogenous free gingival graft (FGG)

ELIGIBILITY:
Inclusion Criteria:

* absence or deficiency of keratinized tissue (< 1mm) in two homologous contralateral sites of inferior premolars
* Miller Class I or II gingival recession
* Absence of radiographic bone loss
* Vital tooth or with adequate endodontic treatment
* Root surfaces without caries
* Good oral hygiene (plaque index < 20%)

Exclusion Criteria:

* Allergic to penicillin
* Presenting systemic disease that impede surgical procedure
* Smokers
* Pregnancy
* Intake of calcium channel blockers that cause gingival augmentation

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 1999-02-01 (Actual); Primary Completion 2017-11-30 (Actual); Study Completion 2017-12-20 (Actual)

PRIMARY OUTCOMES:
keratinized tissue width | 18 years
  Distance from gingival margin to mucogingival junction, measured with a periodontal probe in mm. Ideal if mucosa width is > 5mm.

SECONDARY OUTCOMES:
Probing depth | 18 years
  Distance from gingival margin to bottom of gingival sulcus, measured with a periodontal probe. Ideal if < 2mm.
Attachment level | 18 years
  Distance from cemento-enamel junction to bottom of gingival sulcus, measured with a periodontal probe. Ideal if < 2mm.
Recession depth | 18 years
  Distance from cemento-enamel junction to gingival margin, measured with a periodontal probe. Ideal if = 0mm.

CONTACTS AND LOCATIONS:
Locations (1):
- Bauru School of Dentistry, Bauru, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Cummings LC, Kaldahl WB, Allen EP. Histologic evaluation of autogenous connective tissue and acellular dermal matrix grafts in humans. J Periodontol. 2005 Feb;76(2):178-86. doi: 10.1902/jop.2005.76.2.178. PMID 15974840
- [Background] Agarwal C, Tarun Kumar AB, Mehta DS. Comparative evaluation of free gingival graft and AlloDerm((R)) in enhancing the width of attached gingival: A clinical study. Contemp Clin Dent. 2015 Oct-Dec;6(4):483-8. doi: 10.4103/0976-237X.169838. PMID 26681852